CLINICAL TRIAL: NCT02896127
Title: Randomized, Double-blind, Placebo-controlled, Phase III Multicenter Study of Subcutaneous Secukinumab to Compare Efficacy at 16 Weeks With Placebo and Assess Safety and Tolerability up to 52 Weeks in Subjects With Active Ankylosing Spondylitis
Brief Title: Study of Efficacy and Safety of Secukinumab in Patients With Ankylosing Spondylitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2308; 2015-005021-39 (EudraCT Number)
Record Dates: First submitted 2016-05-04; First posted 2016-09-12 (Estimated); Results first posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Ankylosing Spondyloarthritis
Keywords: Ankylosing Spondyloarthritis; Axial spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab (Experimental): Secukinumab 150 mg s.c.
  Arm includes all patients who received at least 1 dose of study drug including placebo switchers at Week 16
  Interventions: Drug: Secukinumab
- Placebo (Placebo Comparator): Placebo s.c.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secukinumab — Induction: 4x 150 mg Secukinumab s.c. weekly
  Maintenance: 150 mg Secukinumab s.c. monthly
  All Subjects received blinded treatment weekly starting at baseline, Weeks 1, 2, 3 and 4, followed by dosing every four weeks starting at Week 4 until Week 16. At Week 16, Group 1 patients continued using secukinumab 150 mg and Group 2 patients started receiving secukinumab 150 mg dosing every four weeks. Treatment was provided open-label from Week 16 onward, as all patients took 150 mg s.c. every 4 weeks; however, subjects, investigators, and site staff remained blinded to initial randomized group assignment.
  Other Names: AIN457
  Arms: Secukinumab
Drug: Placebo — Induction: 4x placebo s.c. weekly Maintenance: placebo s.c. monthly
  Arms: Placebo

SUMMARY:
The purpose of this trial is to demonstrate the clinical efficacy at week 16; and to demonstrate safety and tolerability of secukinumab compared to placebo in patients with ankylosing spondylitis at week 16 and long term safety up to Week 52.

DETAILED DESCRIPTION:
This multicenter study used a randomized, double-blind, placebo-controlled, parallel-group design. A screening period running up to 10 weeks before randomization was used to assess eligibility, followed by 52 weeks of treatment.

At baseline, subjects were randomized to one of the two treatment groups:

* Group 1: 300 subjects, secukinumab 150 mg (1 mL, 150 mg/mL) s.c. pre-filled syringes (PFS) at BSL, Weeks 1, 2, and 3, followed by administration every four weeks starting at Week 4
* Group 2: 150 subjects, placebo (1 mL) s.c. PFS at BSL, Weeks 1, 2, 3, 4, 8, and 12, followed by secukinumab 150 mg (1 mL, 150 mg/mL) administration every four weeks starting at Week 16

The subjects were stratified at randomization according to the region (China and non-China). Approximately 70% of randomized subjects were from China (327 Chinese subjects) in order to evaluate the efficacy and safety in this subject population. No more than 30% TNFα inhibitor inadequate responders (TNF-IR) subjects were to be enrolled in the study.

Starting at Week 16, all subjects switched to open-label secukinumab 150 mg, including all placebo subjects; however, all subjects and investigators/site staff remained blinded to the original randomized treatment group assignment (150 mg vs placebo). Study treatment continued up to Week 48.

An end of treatment visit was done 4 weeks after last study treatment administration and a post treatment follow-up visit was done 12 weeks after last study treatment administration for all subjects (regardless of whether they completed the entire study as planned or discontinued prematurely).

Subjects were instructed in detail how to self-administer the s.c. injection using PFS. Each injection was administered into an appropriate injection site of the body (thighs, arms, or abdomen). All injections were performed at the study site. Site personnel administered the injections to subjects who were not able to, or felt insecure to self-administer. Rescue medication was not allowed until Week 20. However, subjects who were deemed by the investigator not to be benefiting from the study treatment based on safety and efficacy assessments or for any reason of their own accord were free to discontinue participation in the study at any time.

ELIGIBILITY:
Inclusion Criteria:

Male or non-pregnant, non-lactating female patients at least 18 years of age

Diagnosis of moderate to severe AS with prior documented radiologic evidence (x-ray or radiologist's report) fulfilling the Modified New York criteria for AS:

* Active AS assessed by BASDAI ≥4 (0-10) at Baseline
* Spinal pain as measured by BASDAI question #2 ≥ 4 cm (0-10 cm) at Baseline
* Total back pain as measured by VAS ≥ 40 mm (0-100 mm) at Baseline Patients should have had inadequate response or failure to respond to at least 2 NSAIDs at an approved dose for a minimum of 4 weeks in total and a minimum of 2 weeks for each NSAID prior to randomization, or less than 4 weeks if therapy had to be withdrawn due to intolerance, toxicity or contraindications Patients who are regularly taking NSAIDs (including COX-1 or COX-2 inhibitors) as part of their AS therapy are required to be on a stable dose for at least 2 weeks before randomisation Patients who have been on a TNFα inhibitor (not more than one) must have experienced an inadequate response to previous or current treatment given at an approved dose for at least 3 months prior to randomization or have been intolerant to at least one administration of an anti-TNFα agent

Exclusion Criteria:

* Chest X-ray or MRI with evidence of ongoing infectious or malignant process

  * Patients taking high potency opioid analgesics
  * Previous exposure to secukinumab or any other biologic drug directly targeting IL-17 or IL-17 receptor
  * Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2019-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- China (17):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Xiamen, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Taiyuan, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Bengbu
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Shanxi Province
  - Novartis Investigative Site, Tianjin
  - Novartis Investigative Site, Zhejiang
  - Novartis Investigative Site, Zhenjiang
- Czechia (4):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště
- South Korea (5):
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
- United Kingdom (9):
  - Novartis Investigative Site, Reading, Berkshire
  - Novartis Investigative Site, Bradford, West Yorkshire
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Doncaster
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Southampton
  - Novartis Investigative Site, Wigan

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Merola JF, McInnes IB, Deodhar AA, Dey AK, Adamstein NH, Quebe-Fehling E, Aassi M, Peine M, Mehta NN. Effect of Secukinumab on Traditional Cardiovascular Risk Factors and Inflammatory Biomarkers: Post Hoc Analyses of Pooled Data Across Three Indications. Rheumatol Ther. 2022 Jun;9(3):935-955. doi: 10.1007/s40744-022-00434-z. Epub 2022 Mar 19. PMID 35305260
- [Derived] van der Horst-Bruinsma I, Miceli-Richard C, Braun J, Marzo-Ortega H, Pavelka K, Kivitz AJ, Deodhar A, Bao W, Porter B, Pournara E. A Pooled Analysis Reporting the Efficacy and Safety of Secukinumab in Male and Female Patients with Ankylosing Spondylitis. Rheumatol Ther. 2021 Dec;8(4):1775-1787. doi: 10.1007/s40744-021-00380-2. Epub 2021 Oct 7. PMID 34618347
- [Derived] Huang F, Sun F, Wan WG, Wu LJ, Dong LL, Zhang X, Kim TH, Sengupta R, Senolt L, Wang Y, Qiu HM, Porter B, Haemmerle S. Secukinumab provided significant and sustained improvement in the signs and symptoms of ankylosing spondylitis: results from the 52-week, Phase III China-centric study, MEASURE 5. Chin Med J (Engl). 2020 Nov 5;133(21):2521-2531. doi: 10.1097/CM9.0000000000001099. PMID 32925287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The majority of subjects completed 52 weeks of treatment. After Week 16 all participants originally assigned to placebo switched to AIN457 150 mg s.c. Four out of the 153 assigned to the placebo group discontinued before Week 16.
Pre-assignment Details: All patients independent of completer status were asked to enter follow up whenever they exited the study no matter at what time in their participation. Moreover, not all participants who completed Week 52 entered the follow up period and some did not complete follow-up. Therefore, the number of participants who started the follow-up period is not equal to the number of participants who completed the previous period.
Groups:
- Secukinumab: AIN457 150 mg s.c.
Period: COMPLETED WEEK 52
Arm/Group | Secukinumab | Placebo
Started (Started the Week 52 period) | 305 | 153 (Includes participants originally assigned to placebo and switched to AIN457150 mg after Wk 16.)
Completed (Discontinued before or at Week 52) | 278 | 142
Not Completed | 27 | 11
Not completed — Adverse Event | 9 | 2
Not completed — Lack of Efficacy | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Pregnancy | 2 | 0
Not completed — Withdrawal by Subject | 12 | 4
Not completed — Technical problems | 1 | 0
Period: COMPLETED POST-TREATMENT FOLLOW UP
Arm/Group | Secukinumab | Placebo
Started (All patients independent of completer status were asked to enter follow up whenever they exited the study no matter at what time in their participation. Moreover, not all participants who completed Week 52 entered the follow up period and some did not complete follow-up. Therefore, the number of participants who started the follow-up period is not equal to the number of participants who completed the previous period.) | 280 (Participants enter follow-up if they exited before Wk 52 Thus numbers different from previous period) | 139 (Participants enter follow-up if they exited before Wk 52 Thus numbers different from previous period)
Completed | 276 (Participants enter follow-up if they exited before Wk 52 Thus numbers different from previous period) | 134 (Participants enter follow-up if they exited before Wk 52 Thus numbers different from previous period)
Not Completed | 4 | 5
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was comprised of all subjects from the randomized set to whom study treatment had been assigned. Following the intent-to-treat principle, subjects were evaluated according to the treatment assigned to at randomization, but actual stratum, if stratified randomization was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab | Placebo | Total
Number analyzed (Participants) | 305 | 153 | 458
Age, Categorical [Count of Participants; unit: Participants] — mean age in years Population: Randomized Analysis Set
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 303 | 152 | 455
    >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants] — Full analysis set (FAS) Population: FAS
  Participants
    Female | 53 | 21 | 74
    Male | 252 | 132 | 384
Race/Ethnicity, Customized [Number; unit: participants] — Full analysis set (FAS) Population: FAS
  participants
    Asian | 239 | 130 | 369
    White | 64 | 23 | 87
    Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Participants Who Achieve an ASAS 20 Response (Assessment of SpondyloArthritis International Society Criteria)
Description: ASAS20 response is defined as an improvement of ≥20% and ≥1 units on a scale of 10 in at least three of the four ASAS main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain
Time Frame: Week 16
Population: Full Analysis Set (FAS) was comprised of all subjects from the randomized set to whom study treatment had been assigned. Following the intent-to-treat principle, subjects were evaluated according to the treatment assigned to at randomization, but actual stratum, if stratified randomization was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 305 | 153
Participants | 178 | 56
Statistical Analysis 1: Comparison: Secukinumab vs Placebo; Test type: Superiority; p < .0001, Regression, Logistic; Odds Ratio (OR) = 2.47, 95% CI 2-sided [1.65 to 3.69]; PTFU=post-treatment follow-up (12 weeks after last study treatment) 95% confidence intervals are from a score method with continuity correction

2. Secondary Outcome: The Proportion of Participants Who Achieve an ASAS40 Response
Description: ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain
  The number analyzed for some of continuous outcome variables are the number of participants for whom the specific outcome data were available. Thus the number for these variables differs from the FAS.
Time Frame: The secondary outcome analysis occurred only at Week 16. Thus, while data were collected beyond week 16, they were not part of the secondary outcomes.
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 294 | 146
Participants | 138 | 27

3. Secondary Outcome: Change in hsCRP Over Time
Description: hsCRP is measured as a marker of inflammation from blood samples during the study
  The number analyzed for some of continuous outcome variables are the number of participants for whom the specific outcome data were available. Thus the number for these variables differs from the FAS.
Time Frame: Change from baseline to Week 16. The secondary outcome analysis occurred only at Week 16. Thus, while data were collected beyond week 16, they were not part of the secondary outcomes.
Population: FAS
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 295 | 146
mg/l | -11.78 (22.919) | -0.79 (20.023)

4. Secondary Outcome: Percentage of Participants Who Achieve an ASAS 5/6 at Week 16
Description: The ASAS 5/6 improvement criteria is an improvement of ≥20% in at least five of all six domains
  The number analyzed for some of continuous outcome variables are the number of participants for whom the specific outcome data were available. Thus the number for these variables differs from the FAS.
Time Frame: Week 16: The secondary outcome analysis occurred only at Week 16. Thus, while data were collected beyond week 16, they were not part of the secondary outcomes.
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 295 | 146
percentage of participants | 50.5 [44.7 to 56.3] | 19.2 [13.3 to 26.7]

5. Secondary Outcome: Participants With BASDAI Response at 16 Weeks
Description: The BASDAI or Bath Ankylosing Spondylitis Disease Activity Index consists of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which is used to answer 6 questions pertaining to the 5 major symptoms of AS
  The number analyzed for some of continuous outcome variables are the number of participants for whom the specific outcome data were available. Thus the number for these variables differs from the FAS.
Time Frame: as for outcome 2
Population: FAS
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 295 | 149
percent of participants | 41.7 [36.0 to 47.6] | 22.6 [16.3 to 30.4]

6. Secondary Outcome: Change in Short Form (36) - PCS Responders (Improvement of >= 2.5 Points) at Week 16
Description: The Physical Component Summary (PCS) SF-36 is an instrument to measure health-related quality of life among healthy patients and patients with acute and chronic conditions
  The number analyzed for some of continuous outcome variables are the number of participants for whom the specific outcome data were available. Thus the number for these variables differs from the FAS.
Time Frame: as for outcome 2
Population: FAS
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 301 | 149
percent of participants | 71.8 [66.3 to 76.7] | 61.1 [52.7 to 68.8]

7. Secondary Outcome: Change in ASQoL Score Over Time
Description: The Ankylosing Spondylitis Quality of Life (ASQoL) is an instrument to assess health-related quality of life among adult patients with Ankylosing Spondylitis.
  Each statement on the ASQoL is given a score of "1" or "0". A score of "1" is given where the item is affirmed, indicating adverse QoL. All item scores are summed to give a total score or index. Scores can range from 0 (good QoL) to 18 (poor QoL).
Time Frame: change from baseline to Week 16
Population: FAS
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 305 | 153
scores | -4.6 (4.98) | -2.6 (4.28)

8. Secondary Outcome: The Proportion of Patients Who Achieve an ASAS Partial Remission
Description: The The Assessment in SpondyloArthritis International Society (ASAS) partial remission criteria are defined as a value not above 2 units in each of the four main domains on a scale of 10
  The number analyzed for some of continuous outcome variables are the number of participants for whom the specific outcome data were available. Thus the number for these variables differs from the FAS.
Time Frame: Week 16
Population: FAS
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Secukinumab | Placebo
Number analyzed (Participants) | 294 | 146
percent of participants | 17.7 [13.6 to 22.6] | 7.5 [4.0 to 13.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment up to week 52
Description: An adverse event (AE) is any sign or symptom that occurs during the study treatment period. Patients randomized to placebo at baseline are reported under Placebo up for AEs starting before switching to Secukinumab. Starting from Week 16 onwards, all patients on placebo still in the study were re-assigned to secukinumab and AEs starting after this switch will be counted in the Any AIN457 150 mg group.
Groups:
- Any AIN457 150 mg: This arm includes all patients who received at least 1 dose of study drug.
- Placebo: All patients randomized to placebo from baseline up to week 16.
Arm/Group | Any AIN457 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/453 | 0/153
Serious Adverse Events (participants affected / at risk) | 33/453 | 3/153
Other Adverse Events (participants affected / at risk) | 282/453 | 60/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=453) | Placebo (N=153)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Bronchogenic cyst (Congenital, familial and genetic disorders) | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Iridocyclitis (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Appendix disorder (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Anal abscess (Infections and infestations) | 3 | 0
Appendicitis (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 1 | 0
Pneumonia mycoplasmal (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Electric injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular injury (Injury, poisoning and procedural complications) | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0
Optic neuritis (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 0
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=453) | Placebo (N=153)
Abdominal discomfort (Gastrointestinal disorders) | 15 | 1
Diarrhoea (Gastrointestinal disorders) | 35 | 6
Mouth ulceration (Gastrointestinal disorders) | 18 | 2
Fatigue (General disorders) | 12 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 24 | 3
Nasopharyngitis (Infections and infestations) | 46 | 10
Pharyngitis (Infections and infestations) | 14 | 1
Upper respiratory tract infection (Infections and infestations) | 145 | 29
Urinary tract infection (Infections and infestations) | 16 | 5
Alanine aminotransferase increased (Investigations) | 24 | 3
Aspartate aminotransferase increased (Investigations) | 10 | 2
Protein urine present (Investigations) | 11 | 0
White blood cell count decreased (Investigations) | 17 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 12 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 26 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Dizziness (Nervous system disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 | 2
Rash (Skin and subcutaneous tissue disorders) | 10 | 0
Hypertension (Vascular disorders) | 11 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT02896127/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT02896127/SAP_001.pdf